CLINICAL TRIAL: NCT03261544
Title: Abductor Reattachment Methods in Proximal Femur Replacements: What is the Best Method?
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00082717
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Sarcoma; Bone Metastases; Proximal Femur Replacement
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Proximal Femur Replacement: The proximal femur is a common site for primary bone sarcomas and metastatic disease. The purpose of this study is to assess the functional outcomes in patients undergoing proximal femur resection and reconstruction with an endoprosthesis, based on the abductor muscle repair technique.
  Interventions: Procedure: Proximal Femur Replacement

INTERVENTIONS:
Procedure: Proximal Femur Replacement — The purpose of this study is to assess the functional outcomes in patients undergoing proximal femur resection and reconstruction with an endoprosthesis, based on the abductor muscle repair technique.

SUMMARY:
The purpose of this study is to assess the functional outcomes in patients undergoing proximal femur resection and reconstruction with an endoprosthesis, based on the abductor muscle repair technique. The investigators hypothesize that those patients who receive reattachment of the abductors directly into the prosthesis will have better functional outcomes overall. Furthermore, the investigators plan to develop a simple, cost effective, and reproducible method to assess abductor function at clinical post-operative visits through plain radiographs.

DETAILED DESCRIPTION:
Patients treated for proximal femur replacements at Duke University Medical Center by Orthopaedic Oncology trained surgeons. The Duke DEDUCE database will be used to identify retrospective patients using the above mentioned CPT codes. Individual chart review of the electronic medical record will then be used to identify those receiving a proximal femur replacement. Maximum number of charts to be reviewed in the study will be 300. Of these 300 charts, the investigators plan to consent 25 subjects who have return appointments scheduled. The investigators also plan to consent 25 preoperative patients, for a total of 50 subjects.

ELIGIBILITY:
Inclusion Criteria:

• Has undergone or is scheduled for proximal femur replacement by an Ortho Oncology surgeon

Exclusion Criteria:

* Non-ambulatory before or after the procedure
* Subjects who, in the opinion of the investigator, have not or likely will not complete at least some portion of the investigator's recommended follow-up

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated for proximal femur replacements at Duke University Medical Center by Orthopaedic Oncology trained surgeons. The Duke DEDUCE database will be used to identify retrospective patients using the above mentioned CPT codes. Individual chart review of the electronic medical record will then be used to identify those receiving a proximal femur replacement. Maximum number of charts to be reviewed in the study will be 300. Of these 300 charts, the investigators plan to consent 25 subjects who have return appointments scheduled. The investigators also plan to consent 25 preoperative patients, for a total of 50 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-11-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
The Musculoskeletal Tumor Society (MSTS) score | up to 24 months postoperatively
  The Musculoskeletal Tumor Society (MSTS) score of extremity function. The total score ranges from 0 to 30, with higher scores indicating better function.
Harris Hip Score | up to 24 months postoperatively
  The Harris Hip Score (HHS) is a clinician-based outcome measure that is frequently used for the evaluation of patients following a Total Hip Arthroplasty (THA). The survey has ten questions and scores ranging from 0-100, with higher scores representing less dysfunction and better outcomes.
Number of patients with an implant-related complication as reported on the adverse event form upon participation completion. | up to 24 months postoperatively
  The adverse event form records the occurence of implant-related complications that occur during study participation.

SECONDARY OUTCOMES:
Gait Analysis as reported on the study's case report form | up to 24 months postoperatively
  Motion data collected from gait analysis testing will be evaluated with OpenCap.

CONTACTS AND LOCATIONS:
Overall Officials: William Eward, MD, DVM, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States